## **Cover Page**

Title: Primary Cecal Pathologies Presenting as Acute Abdomen and Critical Appraisal of Their

Current Management Strategies in Emergency Settings

NCT Identifier Number: Not assigned

**Document Date:** 01/01/2016

## **AIMS & OBJECTIVES**

The objective of this study was to identify the reported causes of cecal pathology presenting as acute abdomen in medical literature and the various causes presenting in our setting, to identify the pattern of common pathologies in our setup, to discuss morbidity and mortality associated with cecal pathologies and to critically analyse the various management modalities commonly employed for cecal pathologies presenting as acute abdomen.

## **MATERIALS & METHODS**

This is a retrospective analysis of the prospectively collected data of patients admitted to our unit in last 10 years for acute abdomen, in whom cecal pathology was identified as the prime culprit.

Inclusion Criteria: All adult patients presenting in emergency department with acute abdomen were included in study in whom cecal pathology as the cause of acute abdomen was suspected clinically and/or on imaging and further confirmed per-operatively and/or on histopathological examination (HPE) or on imaging. Patients identified with primarily a cecal pathology who had acute pain abdomen as the initial symptom but who didn't presented immediately due to various reasons<sup>1</sup> were also included in the study as it is a well-documented fact that patients in developing countries like ours, especially those who live in rural areas or who are illiterate often resort to indigenous methods of treatment or take symptomatic treatment from local practitioners before presenting to a tertiary centre like ours for definitive treatment. Also, only those patients who were operated within 24 hours of index admission in the emergency operation theatre (EOT) by a registrar or faculty member itself after initial resuscitation were included in the study.

Exclusion Criteria: Patients with sub-acute, intermittent or chronic pain; when predominant symptoms were attributable to some other cause even with concomitant presence of a cecal pathology; when predominant pathology was not cecal and patients with cecal pathology operated as an elective case were excluded from our study. Thus patients diagnosed to be having appendiceal stump blowout, perforation of base of appendix, ileocecal tuberculosis or intussusception were not included.

We analysed this data of patients admitted to our unit for acute abdomen in whom cecal pathology was the primary cause for the various management options employed and the final outcome of these patients.